CLINICAL TRIAL: NCT04648956
Title: Cross-cultural Adaptation and Psychometric Properties of the Arabic Version of the Intermittent and Constant Osteoarthritis Pain Questionnaire
Brief Title: Arabic Version of the ICOAP Questionnaire
Status: Completed | Type: Observational
Sponsor: Prince Sultan Military College of Health Sciences (Other)
Collaborators: King Fahd Military Medical Complex (Unknown)
Responsible Party: Principal Investigator, Ahmed Farrag, Assisstant Professor, Prince Sultan Military College of Health Sciences
Other Study IDs: IRB-2020-PT-031
Record Dates: First submitted 2020-11-18; First posted 2020-12-02 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
Keywords: ICOAP questionnaire; Arabic; Cross-Cultural adaptation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee/Hip osteoarthritis: Patients referred for physical therapy rehabilitation
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Standard treatment — Participants shall fill the ICOAP-Ar questionnaire three times within one month in addition to other questionnaires including the KOOS/HOOS, and the Global Rating of Change Scale (GRoC). The first two times will be within a time frame of 48-72 hours. The third time will be after one month.
  Other Names: ICOAP questionnaire

SUMMARY:
A study to translate and cross-culturally adapt the Intermittent and Constant Osteoarthritis Pain (ICOAP) measurement tool into the Arabic language, and assess its psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must meet the knee and hip osteoarthritis (OA) diagnostic criteria according to the American College of Rheumatology (ACR).

Exclusion Criteria:

1. rheumatoid arthritis
2. serious pathological conditions (inflammatory arthritis and malignancy)
3. total or partial arthroplasty of the affected joint
4. individuals who cannot read and understand documents written in the Arabic language.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee/Hip osteoarthritis patients recruited from the local community receiving physical therapy rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Content Validity | 1 day
  Assessed using the Content Validity Index (CVI) with an acceptable value of at least 0.8.
Construct Validity | 1 day
  Assessed by calculating the Spearman's correlation coefficient (ρ) between the Arabic ICOAP (ICOAP-Ar) score and the relevant pain and symptoms score of the Knee Injury and Osteoarthritis Outcome Score (KOOS) and Hip Injury and Osteoarthritis Outcome Score (HOOS) measurement tools. The coefficient is classified as follows: ρ = 0.3-0.7 moderate correlation, and >0.7 strong correlation.
Internal Consistency | 48-72 hours
  Assessed by calculating the Cronbach's alpha (α) and the corrected item-total correlation. A Cronbach's α value of ≥0.7, and corrected item-total correlation, measured using the Pearson correlation coefficient, of ≥0.3 will be considered acceptable.
Test-retest Reliability | 48-72 hours
  Assessed by calculating the intraclass correlation coefficient (ICC) between the ICOAP-Ar scores of the first two test sessions. An ICC value of >0.8, and 0.6-0.8 will be considered as excellent and good correlation, respectively.

SECONDARY OUTCOMES:
Responsiveness | 4 weeks
  Participants will be categorized according to their reported Global Rating of Change (GRoC) Scale scores to either improved (GRoC ≥3) or stable group (GRoC <3 to >-3) and between-group comparison of each group's ICOAP-Ar scores will be performed using unpaired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Farrag, PhD, Principal Investigator — Prince Sultan Military College of Health Sciences
Locations (1):
- Prince Sultan Military College of Health Sciences, Dhahran, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided